CLINICAL TRIAL: NCT03703869
Title: A 12-month Prospective Observational Study Assessing the Real-world Clinical Effectiveness, Safety and Health-economic Benefits of Toujeo® Initiation After Oral Antidiabetic Drug Failure in Insulin-naïve Patients With Type 2 Diabetes Mellitus
Brief Title: Twelve -Month Study Observing How Insulin-naïve Patients With Type 2 Diabetes Mellitus Manage Diabetes Using Toujeo® After Oral Antidiabetic Drug Failure, the Side Effect of Toujeo®, and The Cost.
Acronym: ATOS
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS14708; U1111-1215-0174 (Other: UTN)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Insulin glargine (U300): Insulin glargine (U300) dosage and dosing time as per local product labeling
  Interventions: Drug: Insulin glargine (U300)

INTERVENTIONS:
Drug: Insulin glargine (U300) — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous injection
  Other Names: HOE901, Toujeo, Toujeo Solostar

SUMMARY:
Primary Objective:

Assess effectiveness of insulin glargine (U300) in achieving glycemic goal measured by hemoglobin A1c (HbA1c).

Secondary Objectives:

* Assess effectiveness in achieving glycemic goal measured by HbA1c;
* Assess effectiveness on change in HbA1c, fasting plasma glucose (FPG) and self-monitored plasma glucose (SMPG) ;
* Assess requirement for intensification of therapy by additional antidiabetics.
* Assess incidence of hypoglycemia;
* Assess other safety endpoints: adverse events (AEs), serious adverse events (SAEs);
* Assess change in body weight.

DETAILED DESCRIPTION:
Patients will be observed for one year

ELIGIBILITY:
Inclusion criteria :

* Signed patient informed consent;
* Type 2 diabetes mellitus;
* Treated with at least 1 oral antidiabetic drug (OAD) for at least 6 months;
* Hemoglobin A1c (HbA1c) >7.0 % and ≤11% within 3 months of study baseline;
* Physicians' decision in accordance with the current local guidelines to add basal insulin glargine U300 to an existing OAD regimen

Exclusion criteria:

* Diabetes mellitus other than type 2;
* Contraindication to insulin glargine U300 according to local product labelling;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Insulin-naïve patients with type 2 diabetes mellitus and Oral Antidiabetic Drug failure
Sampling Method: Non-Probability Sample
Enrollment: 4589 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c at month 6 | Baseline, month 6
  Percentage of patients achieving Hemoglobin A1c <7.0%.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline, months 3, 6, 12
  Change from baseline in HbA1c at 3, 6, and 12 months
Change in fasting plasma glucose | Baseline, months 3, 6, 12
  Change from baseline in Fasting Plasma Glucose at 3, 6, and 12 months
Change in Self-Monitored Plasma Glucose | Baseline, months 3, 6, 12
  Change from baseline in Self-Monitored Plasma Glucose at 3, 6, and 12 months
Hypoglycemia | Baseline to month 12
  Number of participants with symptomatic hypoglycemic events
Adverse events | Baseline to month 12
  Number of participants with Adverse Events
Serious adverse events | Baseline to month 12
  Number of participants with Serious Adverse Events
Body weight | Baseline to month 12
  Change in average body weight

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (388):
- Colombia (9):
  - Investigational Site Number 1700001, Barranquilla
  - Investigational Site Number 1700004, Bogotá
  - Investigational Site Number 1700010, Bogotá
  - Investigational Site Number 1700005, Cali
  - Investigational Site Number 1700009, Cali
  - Investigational Site Number 1700003, Ibagué
  - Investigational Site Number 1700007, Manizales
  - Investigational Site Number 1700006, Popayán
  - Investigational Site Number 1700002, Zipaquirá
- Egypt (17):
  - Investigational Site Number 8180017, Al Mansurah
  - Investigational Site Number 8180015, Alexandria
  - Investigational Site Number 8180007, Alexandria
  - Investigational Site Number 8180008, Alexandria
  - Investigational Site Number 8180012, Alexandria
  - Investigational Site Number 8180018, Alexandria
  - Investigational Site Number 8180001, Cairo
  - Investigational Site Number 8180005, Cairo
  - Investigational Site Number 8180006, Cairo
  - Investigational Site Number 8180016, Cairo
  - Investigational Site Number 8180020, Cairo
  - Investigational Site Number 8180003, Giza
  - Investigational Site Number 8180011, Giza
  - Investigational Site Number 8180002, Giza
  - Investigational Site Number 8180009, Giza
  - Investigational Site Number 8180014, Giza
  - Investigational Site Number 8180013, Portsaeid
- India (127):
  - Investigational Site Number 3560056, Ahmedabad
  - Investigational Site Number 3560021, Ahmedabad
  - Investigational Site Number 3560049, Ahmedabad
  - Investigational Site Number 3560077, Ahmedabad
  - Investigational Site Number 3560068, Ahmedabad
  - Investigational Site Number 3560014, Aurangabad
  - Investigational Site Number 3560081, Bangalore
  - Investigational Site Number 3560088, Bangalore
  - Investigational Site Number 3560066, Bangalore
  - Investigational Site Number 3560009, Bangalore
  - Investigational Site Number 3560059, Bangalore
  - Investigational Site Number 3560064, Bangalore
  - Investigational Site Number 3560075, Bangalore
  - Investigational Site Number 3560122, Bangalore
  - Investigational Site Number 3560044, Belagavi
  - Investigational Site Number 3560074, Bengaluru
  - Investigational Site Number 3560046, Bengaluru
  - Investigational Site Number 3560116, Bhabaneswar
  - Investigational Site Number 3560062, Bhubaneswar
  - Investigational Site Number 3560106, Chandigarh
  - Investigational Site Number 3560126, Chandigarh
  - Investigational Site Number 3560110, Chennai
  - Investigational Site Number 3560029, Chennai
  - Investigational Site Number 3560080, Chennai
  - Investigational Site Number 3560067, Chennai
  - Investigational Site Number 3560030, Chennai
  - Investigational Site Number 3560008, Chennai
  - Investigational Site Number 3560031, Chennai
  - Investigational Site Number 3560011, Chennai
  - Investigational Site Number 3560124, Chennai
  - Investigational Site Number 3560105, Chennai
  - Investigational Site Number 3560098, Chennai
  - Investigational Site Number 3560104, Chennai
  - Investigational Site Number 3560133, Chennai
  - Investigational Site Number 3560012, Coimbatore
  - Investigational Site Number 3560131, Coimbatore
  - Investigational Site Number 3560032, Delhi
  - Investigational Site Number 3560041, Delhi
  - Investigational Site Number 3560108, Delhi
  - Investigational Site Number 3560002, Delhi
  - Investigational Site Number 3560019, Delhi
  - Investigational Site Number 3560047, Delhi
  - Investigational Site Number 3560102, Delhi
  - Investigational Site Number 3560020, Delhi
  - Investigational Site Number 3560085, Delhi
  - Investigational Site Number 3560118, Erode
  - Investigational Site Number 3560051, Guwahati
  - Investigational Site Number 3560094, Guwahati
  - Investigational Site Number 3560087, Guwahati
  - Investigational Site Number 3560113, Guwahati
  - Investigational Site Number 3560070, Guwahati
  - Investigational Site Number 3560097, Guwahati
  - Investigational Site Number 3560109, Gwalior
  - Investigational Site Number 3560089, Haryāna
  - Investigational Site Number 3560135, Howrah
  - Investigational Site Number 3560096, Howrah
  - Investigational Site Number 3560045, Hyderabad
  - Investigational Site Number 3560058, Hyderabad
  - Investigational Site Number 3560036, Hyderabad
  - Investigational Site Number 3560069, Hyderabad
  - Investigational Site Number 3560035, Hyderabad
  - Investigational Site Number 3560024, Hyderabad
  - Investigational Site Number 3560027, Hyderabad
  - Investigational Site Number 3560043, Hyderabad
  - Investigational Site Number 3560100, Hyderabad
  - Investigational Site Number 3560107, Hyderabad
  - Investigational Site Number 3560034, Hyderabd
  - Investigational Site Number 3560111, Jaipur
  - Investigational Site Number 3560123, Jaipur
  - Investigational Site Number 3560134, Jaipur
  - Investigational Site Number 3560017, Jaipur
  - Investigational Site Number 3560022, Jaipur
  - Investigational Site Number 3560073, Jalandhar
  - Investigational Site Number 3560005, Kanpur
  - Investigational Site Number 3560125, Kanpur
  - Investigational Site Number 3560026, Kochi
  - Investigational Site Number 3560018, Kochi
  - Investigational Site Number 3560050, Kochi
  - Investigational Site Number 3560016, Kochi
  - Investigational Site Number 3560091, Kolkata
  - Investigational Site Number 3560083, Kolkata
  - Investigational Site Number 3560090, Kolkata
  - Investigational Site Number 3560092, Kolkata
  - Investigational Site Number 3560093, Kolkata
  - Investigational Site Number 3560099, Kolkata
  - Investigational Site Number 3560115, Kolkata
  - Investigational Site Number 3560120, Kolkata
  - Investigational Site Number 3560129, Kolkata
  - Investigational Site Number 3560130, Kolkata
  - Investigational Site Number 3650120, Kolkata
  - Investigational Site Number 3560103, Lucknow
  - Investigational Site Number 3560117, Madurai
  - Investigational Site Number 3560033, Mumbai
  - Investigational Site Number 3560121, Mumbai
  - Investigational Site Number 3560136, Mumbai
  - Investigational Site Number 3560042, Mumbai
  - Investigational Site Number 3560065, Mumbai
  - Investigational Site Number 3560015, Mumbai
  - Investigational Site Number 3560079, Mumbai
  - Investigational Site Number 3560003, Mumbai
  - Investigational Site Number 3560023, Mumbai
  - Investigational Site Number 3560040, Mumbai
  - Investigational Site Number 3560119, Mumbai
  - Investigational Site Number 3560112, Navi Mumbai
  - Investigational Site Number 3560010, Nellore
  - Investigational Site Number 3560086, Noida
  - Investigational Site Number 3560132, Noida
  - Investigational Site Number 3560053, Puducherry
  - Investigational Site Number 3560004, Pune
  - Investigational Site Number 3560038, Pune
  - Investigational Site Number 3560055, Pune
  - Investigational Site Number 3560060, Pune
  - Investigational Site Number 3560072, Rajahmundry
  - Investigational Site Number 3560025, Rajkot
  - Investigational Site Number 3560076, Rajkot
  - Investigational Site Number 3560063, Surat
  - Investigational Site Number 3560084, Tinsukia
  - Investigational Site Number 3560006, Trichy
  - Investigational Site Number 3560001, Trichy
  - Investigational Site Number 3560101, Trichy
  - Investigational Site Number 3560114, Tripura
  - Investigational Site Number 3560039, Trivandrum
  - Investigational Site Number 3560013, Trivandrum
  - Investigational Site Number 3560127, Vijayawada
  - Investigational Site Number 3560061, Visakhapatnam
  - Investigational Site Number 3560054, Visakhapatnam
  - Investigational Site Number 3560128, Yamuna Nagar
- Indonesia (3):
  - Investigational Site Number 3600003, Denpasar
  - Investigational Site Number 3600001, Jakarta
  - Investigational Site Number 3600002, Jakarta
- Israel (5):
  - Investigational Site Number 3760001, Haifa
  - Investigational Site Number 3760002, Petah Tikva
  - Investigational Site Number 3760005, Rishon LeZiyyon
  - Investigational Site Number 3760003, Tel Aviv
  - Investigational Site Number 3760004, Tel Aviv
- Jordan (7):
  - Investigational Site Number 4000002, Amman
  - Investigational Site Number 4000005, Amman
  - Investigational Site Number 4000006, Amman
  - Investigational Site Number 4000008, Amman
  - Investigational Site Number 0004, Amman
  - Investigational Site Number 4000009, Amman
  - Investigational Site Number 0007, Irbid
- Kuwait (8):
  - Investigational Site Number 4140001, Al Jabriya
  - Investigational Site Number 4140010, Al Jabriya
  - Investigational Site Number 4140003, Kuwait City
  - Investigational Site Number 4140004, Kuwait City
  - Investigational Site Number 4140006, Kuwait City
  - Investigational Site Number 4140009, Kuwait City
  - Investigational Site Number 4140011, Kuwait City
  - Investigational Site Number 4140012, Kuwait City
- Lebanon (18):
  - Investigational Site Number 4220017, Airport Road
  - Investigational Site Number 4220008, Aley
  - Investigational Site Number 4220001, Beirut
  - Investigational Site Number 4220015, Beirut
  - Investigational Site Number 4220012, Bir Al Abed
  - Investigational Site Number 4220007, Chtoura
  - Investigational Site Number 4220011, Corniche El Mazraa
  - Investigational Site Number 4220006, El Achrafiyé
  - Investigational Site Number 4220016, El Achrafiyé
  - Investigational Site Number 4220018, Hadath
  - Investigational Site Number 4220013, Hamra
  - Investigational Site Number 4220019, Jal El Baher
  - Investigational Site Number 4220014, Jounieh
  - Investigational Site Number 4220010, Metn
  - Investigational Site Number 4220004, Mount Lebanon
  - Investigational Site Number 4220005, Saida
  - Investigational Site Number 4220003, Sarba
  - Investigational Site Number 4220009, Tyre
- Mexico (10):
  - Investigational Site Number 4840001, Aguascalientes
  - Investigational Site Number 4840009, Celaya
  - Investigational Site Number 4840008, Chihuahua City
  - Investigational Site Number 4840004, Cuernavaca
  - Investigational Site Number 4840007, Durango
  - Investigational Site Number 4840006, Guadalajara
  - Investigational Site Number 4840003, Guadalajara
  - Investigational Site Number 4840005, México
  - Investigational Site Number 4840010, México
  - Investigational Site Number 4840002, México
- Peru (3):
  - Investigational Site Number 6040003, Arequipa
  - Investigational Site Number 6040001, Lima
  - Investigational Site Number 6040002, Lima
- Investigational Site Number 6080001, Dasmarinas Cavite, Philippines
- Russia (125):
  - Investigational Site Number 6430108, Anapa
  - Investigational Site Number 6430170, Arkhangelsk
  - Investigational Site Number 6430171, Arkhangelsk
  - Investigational Site Number 6430172, Arkhangelsk
  - Investigational Site Number 6430019, Astrakhan
  - Investigational Site Number 6430010, Barnaul
  - Investigational Site Number 6430138, Barnaul
  - Investigational Site Number 6430081, Barnaul
  - Investigational Site Number 6430182, Barnaul
  - Investigational Site Number 6430160, Barnaul
  - Investigational Site Number 6430181, Barnaul
  - Investigational Site Number 6430157, Belorechensk
  - Investigational Site Number 6430156, Bryansk
  - Investigational Site Number 6430060, Chaltyr
  - Investigational Site Number 6430087, Cheboksary
  - Investigational Site Number 6430097, Chelyabinsk
  - Investigational Site Number 6430036, Chelyabinsk
  - Investigational Site Number 6430092, Chelyabinsk
  - Investigational Site Number 6430107, Chelyabinsk
  - Investigational Site Number 6430111, Gorodets
  - Investigational Site Number 6430012, Kazan'
  - Investigational Site Number 6430184, Kazan'
  - Investigational Site Number 6430011, Kemerovo
  - Investigational Site Number 6430109, Kemerovo
  - Investigational Site Number 6430072, Kemerovo
  - Investigational Site Number 6430125, Kolomna
  - Investigational Site Number 6430143, Krasnodar
  - Investigational Site Number 6430047, Krasnodar
  - Investigational Site Number 6430136, Krasnodar
  - Investigational Site Number 6430083, Krasnodar
  - Investigational Site Number 6430140, Krasnodar
  - Investigational Site Number 6430021, Krasnodar
  - Investigational Site Number 6430115, Krasnoyarsk
  - Investigational Site Number 6430004, Krasnoyarsk
  - Investigational Site Number 6430068, Lipetsk
  - Investigational Site Number 6430067, Lipetsk
  - Investigational Site Number 6430024, Livny
  - Investigational Site Number 6430128, Moscow
  - Investigational Site Number 6430168, Moscow
  - Investigational Site Number 6430064, Moscow
  - Investigational Site Number 6430065, Moscow
  - Investigational Site Number 6430148, Moscow
  - Investigational Site Number 6430079, Moscow
  - Investigational Site Number 6430101, Moscow
  - Investigational Site Number 6430100, Moscow
  - Investigational Site Number 6430120, Moscow
  - Investigational Site Number 6430130, Moscow
  - Investigational Site Number 6430026, Moscow
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430017, Moscow
  - Investigational Site Number 6430027, Moscow
  - Investigational Site Number 6430057, Moscow
  - Investigational Site Number 6430035, Moscow
  - Investigational Site Number 6430118, Moscow
  - Investigational Site Number 6430146, Moscow
  - Investigational Site Number 6430147, Moscow
  - Investigational Site Number 6430051, Moscow
  - Investigational Site Number 6430149, Moscow
  - Investigational Site Number 6430132, Nizhny Novgorod
  - Investigational Site Number 6430066, Nizhny Novgorod
  - Investigational Site Number 6430129, Nizhny Novgorod
  - Investigational Site Number 6430110, Novomoskovsk
  - Investigational Site Number 6430007, Novosibirsk
  - Investigational Site Number 6430061, Novosibirsk
  - Investigational Site Number 6430023, Novosibirsk
  - Investigational Site Number 6430117, Omsk
  - Investigational Site Number 6430014, Orenburg
  - Investigational Site Number 6430112, Oryol
  - Investigational Site Number 6430137, Oryol
  - Investigational Site Number 6430039, Penza
  - Investigational Site Number 6430164, Penza
  - Investigational Site Number 6430126, Perm
  - Investigational Site Number 6430040, Petrozavodsk
  - Investigational Site Number 6430054, Petrozavodsk
  - Investigational Site Number 6430084, Petrozavodsk
  - Investigational Site Number 6430038, Pushkin
  - Investigational Site Number 6430151, Rostov-on-Don
  - Investigational Site Number 6430090, Rostov-on-Don
  - Investigational Site Number 6430037, Rybinsk
  - Investigational Site Number 6430086, Saint Petersburg
  - Investigational Site Number 6430139, Saint Petersburg
  - Investigational Site Number 6430022, Saint Petersburg
  - Investigational Site Number 6430070, Saint Petersburg
  - Investigational Site Number 643085, Saint Petersburg
  - Investigational Site Number 6430028, Saint Petersburg
  - Investigational Site Number 6430074, Saint Petersburg
  - Investigational Site Number 6430135, Saint Petersburg
  - Investigational Site Number 6430150, Saint Petersburg
  - Investigational Site Number 6430095, Saint Petersburg
  - Investigational Site Number 6430032, Saint Petersburg
  - Investigational Site Number 6430144, Saint Petersburg
  - Investigational Site Number 6430031, Saint Petersburg
  - Investigational Site Number 6430099, Saint Petersburg
  - Investigational Site Number 6430131, Saint Petersburg
  - Investigational Site Number 6430163, Saint Petersburg
  - Investigational Site Number 6430152, Saint Petersburg
  - Investigational Site Number 6430073, Sal'sk
  - Investigational Site Number 6430177, Samara
  - Investigational Site Number 6430046, Samara
  - Investigational Site Number 6430029, Shatura
  - Investigational Site Number 6430155, Smolensk
  - Investigational Site Number 6430121, Smolensk
  - Investigational Site Number 6430089, Sochi
  - Investigational Site Number 6430044, Stavropol
  - Investigational Site Number 6430134, Stavropol
  - Investigational Site Number 6430153, Stavropol
  - Investigational Site Number 6430076, Tambov
  - Investigational Site Number 6430142, Tambov
  - Investigational Site Number 6430013, Tolyatti
  - Investigational Site Number 6430058, Tomsk
  - Investigational Site Number 6430030, Tver'
  - Investigational Site Number 6430169, Tver'
  - Investigational Site Number 6430166, Tver'
  - Investigational Site Number 6430123, Tyumen
  - Investigational Site Number 6430098, Tyumen
  - Investigational Site Number 6430078, Tyumen
  - Investigational Site Number 6430189, Ufa
  - Investigational Site Number 6430041, Ulyanovsk
  - Investigational Site Number 6430114, Vladimir
  - Investigational Site Number 6430018, Volgograd
  - Investigational Site Number 6430052, Vsevolozhsk
  - Investigational Site Number 6430008, Vyksa
  - Investigational Site Number 6430055, Yaroslavl
  - Investigational Site Number 6430033, Yartsevo
  - Investigational Site Number 6430006, Yoshkar-Ola
- Saudi Arabia (8):
  - Investigational Site Number 6820009, Al Ehsa
  - Investigational Site Number 6820006, Jeddah
  - Investigational Site Number 6820001, Jeddah
  - Investigational Site Number 6820008, Jeddah
  - Investigational Site Number 6820010, Jeddah
  - Investigational Site Number 6820007, Jubail
  - Investigational Site Number 6820004, Najrān
  - Investigational Site Number 6820003, Riyadh
- Investigational Site Number 7020001, Singapore, Singapore
- Taiwan (6):
  - Investigational Site Number 1580007, Changhua
  - Investigational Site Number 1580005, Kaohsiung Hsien,
  - Investigational Site Number 1580003, New Taipei City
  - Investigational Site Number 1580004, Taichung
  - Investigational Site Number 1580002, Tainan
  - Investigational Site Number 1580006, Taipei
- Thailand (2):
  - Investigational Site Number 7640002, Bangkok
  - Investigational Site Number 7640001, Bangkok
- Ukraine (20):
  - Investigational Site Number 8040020, Cherkasy
  - Investigational Site Number 8040002, Chernivtsi
  - Investigational Site Number 8040006, Dnipro
  - Investigational Site Number 8040014, Dnipro
  - Investigational Site Number 8040010, Ivano-Frankivsk
  - Investigational Site Number 8040013, Kharkiv
  - Investigational Site Number 8040016, Kharkiv
  - Investigational Site Number 8040001, Kharkiv
  - Investigational Site Number 8040012, Khmelnytskyi
  - Investigational Site Number 8040019, Kyiv
  - Investigational Site Number 8040005, Kyiv
  - Investigational Site Number 8040008, Kyiv
  - Investigational Site Number 8040011, Kyiv
  - Investigational Site Number 8040017, Kyiv
  - Investigational Site Number 8040007, Poltava
  - Investigational Site Number 8040004, Sumy
  - Investigational Site Number 8040009, Ternopil
  - Investigational Site Number 8040018, Ternopil
  - Investigational Site Number 8040003, Vinnytsia
  - Investigational Site Number 8040015, Zaporizhzhia
- United Arab Emirates (18):
  - Investigational Site Number 7840017, Abu Dhabi
  - Investigational Site Number 7840018, Abu Dhabi
  - Investigational Site Number 7840007, Ajman
  - Investigational Site Number 7840001, Dubai
  - Investigational Site Number 7840002, Dubai
  - Investigational Site Number 7840003, Dubai
  - Investigational Site Number 7840004, Dubai
  - Investigational Site Number 7840005, Dubai
  - Investigational Site Number 7840008, Dubai
  - Investigational Site Number 7840009, Dubai
  - Investigational Site Number 7840010, Dubai
  - Investigational Site Number 7840012, Dubai
  - Investigational Site Number 7840013, Dubai
  - Investigational Site Number 7840014, Dubai
  - Investigational Site Number 7840015, Dubai
  - Investigational Site Number 7840016, Dubai
  - Investigational Site Number 7840019, Umm Al Quwain City
  - Investigational Site Number 7840020, Umm Al Quwain City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Tirosh A, Khan N, Vargas-Uricoechea H, Galstyan G, Al Shaikh AR, Makkar BM, Mabunay MA, Melas-Melt L, Pilorget V, Karalliedde J. Effectiveness and Safety of Insulin Glargine 300 U/ml in High-Risk Subgroups (Renal Impairment and Older Age >/= 70 years) of Insulin-Naive People with Type 2 Diabetes: A Post hoc Analysis of Real-World ATOS Study. Diabetes Ther. 2025 Oct;16(10):2045-2061. doi: 10.1007/s13300-025-01785-w. Epub 2025 Sep 8. PMID 40920273
- [Derived] Khan NE, Al Shaikh AAM, Hassoun AAK, Hassan AM, Salah MM, Al Abdella NA, Safarini SSM, Al Dahi WA, Akil YA. Real-World Study on Effectiveness of Insulin Glargine U300 After Oral Antidiabetic Drug Failure in Patients with Type 2 Diabetes in the Gulf Region. Diabetes Ther. 2024 Mar;15(3):691-704. doi: 10.1007/s13300-024-01537-2. Epub 2024 Feb 15. PMID 38355814
- [Derived] Galstyan GR, Tirosh A, Vargas-Uricoechea H, Mabunay MA, Coudert M, Naqvi M, Pilorget V, Khan N. Real-World Effectiveness and Safety of Insulin Glargine 300 U/mL in Insulin-Naive People with Type 2 Diabetes: the ATOS Study. Diabetes Ther. 2022 Jun;13(6):1187-1202. doi: 10.1007/s13300-022-01266-4. Epub 2022 May 9. PMID 35532858